CLINICAL TRIAL: NCT02774811
Title: Primary Glaucoma Treatment Trial in Kenya and South Africa - SLT vs. Medication
Acronym: SLT/med
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to maintain a functional laser in the environment
Sponsor: University College, London (Other)
Collaborators: University of KwaZulu (Other); Kisii Eye Hospital Kisii Kenya (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0167
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Prostaglandins, Synthetic; Bimatoprost; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selective laser trabeculoplasty (Active Comparator): Selective laser trabeculoplasty
  Interventions: Procedure: Selective laser trabeculoplasy; Device: laser
- Prostaglandin analogue (Active Comparator): Prostaglandin analogue topical medical therapy
  Interventions: Drug: Prostaglandin analogue

INTERVENTIONS:
Drug: Prostaglandin analogue — Topical therapy
  Other Names: Bimatoprost
  Arms: Prostaglandin analogue
Procedure: Selective laser trabeculoplasy — Laser therapy into drainage angle
  Arms: Selective laser trabeculoplasty
Device: laser
  Arms: Selective laser trabeculoplasty

SUMMARY:
Multi-centre randomised controlled trial of selective laser trabeculoplasty compared with prostaglandin analogue therapy as primary treatment for high tension open angle glaucoma.

Participating centres are:

Institute of Ophthalmology, UCL, London, UK McCord Hospital, Durban, South Africa Innovation Eye Centre, Kisii, Kenya

DETAILED DESCRIPTION:
A debate continues concerning best first-line therapy for African primary open angle glaucoma. Most African practitioners advocate first line trabeculectomy surgery yet most frequently practice first line drug therapy because of patient acceptance and other issues. In the developed world a range of first line therapies including drug, SLT, cyclodiode ciliary body ablation, trabeculectomy surgery, drainage tube surgery and other drainage procedures (viscocanalostomy, non-penetrating surgery etc) have been advocated.

There is a paucity of good evidence concerning the relative merits of these approaches in an African context. The purpose of this study is to compare two approaches to first line therapy of primary open angle glaucoma in an African population.

Design A two centre randomised prospective trial of SLT vs. prostaglandin analogue first line therapy for primary open angle glaucoma.

Methods African patients with established or newly diagnosed primary open angle glaucoma or patients with POAG currently on single drug therapy (excluding prostaglandin analogues) and elevated IOP are recruited in Innovation Eye Centre in Kisii, Kenya and McCord Hospital, University of KwaZulu-Natal, Durban, South Africa. While if clinically indicated both eyes will be treated, one eye per patient to be included in the study.

After informed consent all patients undergo a standardised examination to establish baseline ocular function and findings. All patients receive counselling in glaucoma, the disease, what it means and the therapy. The patient is then randomised (randomisation in London, contained in sealed opaque envelopes) to receive SLT or prostaglandin analogue therapy. Every effort is made to follow all patients according to a standardised protocol at a minimum of month 3, month 6 and month 12. All therapeutic failures are followed closely to ascertain further management plans and subsequent therapeutic compliance. Follow-up is offered beyond 12 months.

Medical therapy Those randomised to medical therapy patients receive free Prostaglandin analogue in KZN or in Innovation Eye Centre with counselling on drop instillation and instructions for renewal of their prescription. Prescription renewal is to be free of charge.. An appointment is given for review in 3 months. Considerable attention is being paid to estimating compliance including the use of bottle weighing and questionnaires already developed and used locally.

SLT THERAPY Those randomised to SLT will receive counseling on the effects and management of SLT.

System: Selecta II (Lumenis) - Frequency doubled Nd: YAG (532nm) Pre-Laser Treatment

* Topical anesthesia (e.g. proxymetacaine hydrochloride)
* Prophylactic application of alpha agonist or equivalent agent (e.g. brimonidine) to avoid
* Post-op pressure spike

Laser Treatment parameters:

1. Duration 3ns (preset)
2. Spot size 400µ (preset)
3. Number of applications: 100
4. Extent of angle: 360 degree
5. Power (dependent on angle pigmentation)

   * If pigmentation is 1 or 2. start at 0.8 mJ and adjust power in 0.1 mJ increments until visible response (cavitation bubbles - colloquially referred to as "champagne bubbles")
   * If pigment grade is 3 or 4, start at lower energy 0.4 mJ and adjust power in 0.1 mJ increments until visible response
   * When reaching the treatment endpoint (cavitation bubbles), scale down the energy level by 0.1 mJ and remain on that threshold throughout treatment
   * It is recommended to re-evaluate threshold following the treatment of each quadrant, due to variations in TM pigmentation to reach treatment endpoint (cavitation bubbles) Post-Laser Treatment
   * Patient's IOP follow up - one hour post treatment
   * NSAIDS up to 2-3 days post-op, or depending on the level of patient discomfort
   * It is not recommended to prescribe steroidal medication as it may potentially interfere with the SLT mechanism of action.

Follow-up At 3 months Patients will have a structured questionnaire relating to any adverse effects from the therapeutic interventions. They will receive an examination of visual function, external ocular structures and intraocular pressure in addition to the optic nerve head.

Those with unacceptable topical/systemic side effects and those with partial or complete failure of IOP control (see outcomes) will have secondary therapy commenced in the form of timolol 0.5% or, if contraindicated, either brimonidine or oral acetazolamide)). The secondary therapy will either replace or be additive to the primary therapy depending on the initial response.

At 6 months Patients will have a structured questionnaire relating to any adverse effects from therapeutic interventions. They will receive and examination of visual function, external ocular stuctures and intraocular pressure in addition to the optic nerve head.

Those with unacceptable topical/systemic side effects and those with partial or complete failure of IOP control (see outcomes) will have secondary or tertiary therapy commenced in the form of timolol 0.5% or, if contraindicated, either brimonidine or oral acetazolamide)) or surgical intervention in the form of a trabeculectomy with cytotoxic.

At 12 months Patients will have a structured questionnaire relating to any adverse effects from therapeutic interventions. This questionnaire will also include questions relating to their acceptance of the therapy and view of the therapy. They will receive a detailed examination of visual function and ocular parameters.

Those with unacceptable topical/systemic side effects and those with partial or complete failure of IOP control (see outcomes) and those with evidence of glaucoma progression will have secondary or tertiary therapy commenced in the form of timolol 0.5% or, if contraindicated, either brimonidine or oral acetazolamide)) or surgical intervention in the form of a trabeculectomy with cytotoxic.

ELIGIBILITY:
Inclusion Criteria:

* • Consent to inclusion and participation in trial.

  * Characteristic glaucomatous changes in the optic disc. The presence of a focal or diffuse area of optic disc rim loss, so that the neuroretinal rim tissue in any quadrant is less than 5% of the disc diameter in that meridian. Extensive loss of neuroretinal rim tissue with marked optic disc cupping giving a cup disc ratio greater than 0.6.
  * A measured intraocular pressure greater than or equal to 21 mmHg and less than or equal to 30mmHg on at least one visit before the time of entry into the study as measured by Goldmann applanation tonometry.
  * Adequate visualization of angle structures (i.e. clear media and cooperative patient)
  * Black African patients

Exclusion Criteria:

* • Unwillingness to participate in the study

  * Inability/unwillingness to give informed consent
  * Unwillingness to accept randomisation
  * Patient less than 20 years of age
  * Anterior segment neovascularisation
  * Past trauma to the eye or ocular adnexae
  * Retinal or optic nerve neovascularisation
  * Aphakia or pseudophakia
  * Previous ocular surgery Evidence of ocular disease other than glaucoma that might affect the measurements of IOP, assessment of visual function, visual field testing would likely require cataract surgery within 12 months of randomization on systemic medications known to -IOP (e.g. steroids) Pregnancy or female of childbearing age who may be pregnant at time of treatment (LMP).
  * Anyone who is not Black African race

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure reduction | 1 year
  30% reduction complete 15-29% partial success

SECONDARY OUTCOMES:
Compliance | 1 year
  proportion complying with medical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ian Murdoch, MD FRCOphth, Principal Investigator — UCL
Locations (1):
- Innovation Eye Centre, Kisii, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Once publication accepted data to be shared in normal fashion with publication